CLINICAL TRIAL: NCT03622489
Title: Comparing Protocols for Analgesia Following Elective Cesarean Section
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0022-17-WOMC
Record Dates: First submitted 2018-08-05; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-06

CONDITIONS: Postoperative Pain; Post-Cesarean Section
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Ibuprofen; Dipyrone; Tramadol; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tab ibuprofen + IV acetaminophen (Experimental): All women will receive immediately after surgery, in the recovery room:
  1. IV morphin 5 mg, repeat doses every 10 minutes for VNS>3
  2. IV Tramal 100 mg, once
  After Admitted to Maternity ward:
  - Scheduled doses: 08:00 hr, Tab. Ibuprofen 400 mg, and IV Acetaminophen 1 gr 14:00 hr, IV Acetaminophen 1 gr 19:00 hr, Tab. Ibuprofen 400 mg 00:00 hr, IV Acetaminophen 1 gr
  -Additional analgesia if needed according to VNS scale: PO drops Dipyrone 1 gr, for VNS>4, up to 4 times a day, at least 6 hours between doses.
  Tab Tramadex 100 mg, for VNS>6, or if pain persists for 1 hour after receiving Dipyrone, up to 3 times a day, at least 4 hours between doses.
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen 400 mg; Drug: Tramadol; Drug: Morphine; Drug: Tramal
- Tab Ibuprofen + Tab acetaminophen (Experimental): All women will receive immediately after surgery, in the recovery room:
  1. IV morphin 5 mg, repeat doses every 10 minutes for VNS>3
  2. IV Tramal 100 mg, once
  After Admitted to Maternity ward:
  - Scheduled doses: 08:00 hr, Tab. Ibuprofen 400 mg, and PO Acetaminophen 1 gr 14:00 hr, PO Acetaminophen 1 gr 19:00 hr, Tab. Ibuprofen 400 mg 00:00 hr, PO Acetaminophen 1 gr
  - Additional analgesia if needed according to VNS scale: PO drops Dipyrone 1 gr, for VNS>4, up to 4 times a day, at least 6 hours between doses.
  Tab Tramadex 100 mg, for VNS>6, or if pain persists for 1 hour after receiving Dipyrone, up to 3 times a day, at least 4 hours between doses.
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen 400 mg; Drug: Tramadol; Drug: Morphine; Drug: Tramal
- "On demand" analgesia (Experimental): All women will receive immediately after surgery, in the recovery room:
  1. IV morphin 5 mg, repeat doses every 10 minutes for VNS>3
  2. IV Tramal 100 mg, once
  After Admitted to Mternity ward:
  Will not receive scheduled pain medication, but offered some only upon patients' request according to VNS score:
  * Tab. Acetaminophen 1 gr, for VNS 1-3, up to 4 times a day, at east 6 hours between doses.
  * PO drops Dipyrone 1 gr, for VNS 4-7, or if pain persists for 1 hour after receiving Acetaminophen, up to 4 times a day, at least 6 hours between doses.
  * Tab Ibuprofen 400 mg, for VNS 8-10, or if pain persists for 1 hour after receiving Dipyrone, up to 3 times a day, at least 8 hours between doses.
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen 400 mg; Drug: Dipyrone; Drug: Tramadol; Drug: Morphine; Drug: Tramal

INTERVENTIONS:
Drug: Acetaminophen — mentioned above
Drug: Ibuprofen 400 mg — mentioned above
Drug: Dipyrone — mentioned above
  Arms: "On demand" analgesia
Drug: Tramadol — mentioned above
  Other Names: Tramadex
Drug: Morphine — mentioned above
Drug: Tramal — mentioned above

SUMMARY:
Women undergoing elective cesarian section will be assigned to 3 groups for postoperative analgesia:

1. Scheduled doses of IV acetaminophen + PO Ibuprofen
2. Scheduled doses of PO acetaminophen + PO Ibuprofen
3. "On demand" doses of acetaminophen, dipyrone and ibuprofen.

DETAILED DESCRIPTION:
A prospective randomised trial. Women undergoing elective cesarean section will be randomized to three groups. The treatment will be given for 48 hours after surgery. For evealuating objective pain sensation the investigators will be using the Visual Numerical Score (VNS). Demographic characteristics and information about breastfeeding and medications' side effects, will be reviewed from patients' medical scores.

Exclusion criteria: known allergies to one or more of the studies' drugs, general anesthesia, woman undergoing her 3rd cesarean section or more, elective tubal ligation performed at the time of current cesarean section, contraindication for use of one or more of the studies' drugs.

Number of participants: 120

Treatment:

All women will receive immediately after surgery, in the recovery room:

1. IV morphin 5 mg, repeat doses every 10 minutes for VNS>3
2. IV Tramal 100 mg, once

After Admitted to Mternity ward:

* 1st group will be receiving scheduled doses: 08:00 hr, Tab. Ibuprofen 400 mg, and IV Acetaminophen 1 gr 14:00 hr, IV Acetaminophen 1 gr 19:00 hr, Tab. Ibuprofen 400 mg 00:00 hr, IV Acetaminophen 1 gr
* 2nd group will be receiving scheduled doses: 08:00 hr, Tab. Ibuprofen 400 mg, and PO Acetaminophen 1 gr 14:00 hr, PO Acetaminophen 1 gr 19:00 hr, Tab. Ibuprofen 400 mg 00:00 hr, PO Acetaminophen 1 gr
* 1st+2nd group will be given additional analgesia if needed according to VNS scale: PO drops Dipyrone 1 gr, for VNS>4, up to 4 times a day, at least 6 hours between doses.

Tab Tramadex 100 mg, for VNS>6, or if pain persists for 1 hour after receiving Dipyrone, up to 3 times a day, at least 4 hours between doses.

- 3rd group will not receive scheduled pain medication, but offered some only upon patients' request according to VNS score:

* Tab. Acetaminophen 1 gr, for VNS 1-3, up to 4 times a day, at east 6 hours between doses.
* PO drops Dipyrone 1 gr, for VNS 4-7, or if pain persists for 1 hour after receiving Acetaminophen, up to 4 times a day, at least 6 hours between doses.
* Tab Ibuprofen 400 mg, for VNS 8-10, or if pain persists for 1 hour after receiving Dipyrone, up to 3 times a day, at least 8 hours between doses.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing elective cesarian section

Exclusion Criteria:

* known allergies to one or more of the studies' drugs, general anesthesia, woman undergoing her 3rd cesarean section or more, elective tubal ligation performed at the time of current cesarean section, contraindication for use of one or more of the studies' drugs.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Average pain score 48 hours following surgery: visual numerical scale (VNS) | 48 hours
  Using : visual numerical scale (VNS)

CONTACTS AND LOCATIONS:
Overall Officials: Michal Kovo, MD, Study Chair — Wolfson Medical Center
Locations (1):
- Wolfson medical center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dafna L, Herman HG, Ben-Zvi M, Bustan M, Sasson L, Bar J, Kovo M. Comparison of 3 protocols for analgesia control after cesarean delivery: a randomized controlled trial. Am J Obstet Gynecol MFM. 2019 May;1(2):112-118. doi: 10.1016/j.ajogmf.2019.04.002. Epub 2019 Apr 8. PMID 33345816